CLINICAL TRIAL: NCT01113567
Title: Effect of Lactose in Patients With Chronic Liver Disease and Minimal Hepatic Encephalopathy. Double- Blind, Randomized, Controlled Clinical Trial
Brief Title: Effect of Lactose in Patients With Chronic Liver Disease and Minimal Hepatic Encephalopathy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: erminated [The study was withdrawn because of the reconversion of the hospital to care for patients with COVID19. For this reason, it was not possible to continue recruiting and monitoring patients for this clinical study.]
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Responsible Party: Principal Investigator, Segundo Moran Villota, Asociado B, Coordinación de Investigación en Salud, Mexico
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2010-785-016
Record Dates: First submitted 2010-04-28; First posted 2010-04-30 (Estimated); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Hepatic Encephalopathy; Liver Cirrhosis
Keywords: Hepatic Encephalopathy; Liver Cirrhosis; Disaccharides; Lactose; Quality of Life
MeSH Terms: conditions — Hepatic Encephalopathy; Liver Cirrhosis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diet and lactose-free milk (Placebo Comparator): Lactose-free milk
  Interventions: Dietary Supplement: Lactose-free milk
- Diet and whole milk (Active Comparator): Whole milk with lactose
  Interventions: Dietary Supplement: Whole milk

INTERVENTIONS:
Dietary Supplement: Lactose-free milk — 3.5 g of lactose
  Arms: Diet and lactose-free milk
Dietary Supplement: Whole milk — Whole milk with 24 g lactose
  Arms: Diet and whole milk

SUMMARY:
Two groups of patients with minimal hepatic encephalopathy will be studied. The treatment group (n=17) will receive whole milk (24 g lactose) and the control group (n=17) will receive "lactose-free" milk (3.5 g of lactose) two times a day for 21 days. Clinical history, nutritional assessment, biochemical studies, psychometric tests, critical flicker frequency and a quality of life questionnaire will be performed. The patient will be assessed weekly 21 days. An external monitor will control the randomization process in order to allocate the patients into both study group and will not share the assignation codes with anyone until the end of the study.

DETAILED DESCRIPTION:
Mortality due to chronic liver disease is among the first five causes of mortality related to digestive tract and liver diseases in patients on productive age. One of the most frequent complications of chronic liver insufficiency is minimal hepatic encephalopathy (MHE), which affects the quality of life and predisposes to the development of clinical hepatic encephalopathy. There are few evidences on the therapeutic alternatives for minimal hepatic encephalopathy. The administration of non-absorbable disaccharides has been proven to ameliorate MHE. Lactose maldigestion may justify the use of lactose in patients with chronic liver disease as a non-absorbable disaccharide for the treatment of MHE.

The aim of our study is to evaluate the efficacy of lactose administration in patients with minimal hepatic encephalopathy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic liver disease of whichever etiology
* Minimal hepatic encephalopathy
* Lactose maldigestion

Exclusion Criteria:

* Patients with clinical manifestations of hepatic encephalopathy
* Recent use of antibiotics or psychotropic drugs
* Recent use of alcohol abuse
* Gastrointestinal bleeding
* Others neurological disorders that affect the psychometric test
* Chronic renal failure
* Congestive heart failure
* Chronic Obstructive Pulmonary Disease
* Severe symptoms of lactose intolerance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2010-07 (Actual); Primary Completion 2021-07-26 (Actual); Study Completion 2021-07-26 (Actual)

PRIMARY OUTCOMES:
Reversion of Minimal Hepatic Encephalopathy (MHE) in patients with cirrosis | 30 days after intervention
  Improve in Psychometric Hepatic Encephalopathy Score (PHES). The PHES includes five psychometric test: number connectiontests A and B; the digit symbol test; the line tracing test and the serial dotting test. To calculate th PHES, the validated equations for Mexican population will be used. Patients will be diagnosed with MHE when the PHES will be less than -4 points.

SECONDARY OUTCOMES:
Quality of life in patients with cirrhosis and minimal hepatic encephalopathy | 30 days after intervention
  Analyze the number of patients who improve the record of quality of life, that will be evaluated with the Chronic Liver Disease Questionnaire (CLDQ). The score of the six domains and the overall CLDQ was calculated with answers presented on a 7-point likert scale, where number 1 referred to the maximum frequency (always) and 7 to the lowest frequency (never). A change of 0.5 on the 1-7 scale aproximates the important difference in questionnaire score.

CONTACTS AND LOCATIONS:
Overall Officials: Segundo Moran, MD, Principal Investigator — Instituto Mexicano del Seguro Social
Locations (1):
- Instituto Mexicano del Seguro Social, Mexico City, Mexico City, Mexico

REFERENCES:
- See also: Instituto Mexicano del Seguro Social — http://www.imss.gob.mx